CLINICAL TRIAL: NCT04164784
Title: Evaluate the Effect of "Therapeutic Monitoring"（Flash Continuous Glucose Monitoring System）on Blood Glucose Control in Type 2 Diabetes
Brief Title: Effect of "Therapeutic Monitoring" on Blood Glucose Control in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ruijin-20191101
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- therapeutic monitoring (Experimental): Based on the dietary habits from guidelines, the patients will be instructed to adjust the diet according to the ambulatory glucose profile (AGP) and the recorded log monitored by the continuous glucose monitoring system, thereby implementing"therapeutic monitoring".
  Interventions: Behavioral: therapeutic monitoring
- The control group (No Intervention): Patients will be given the basic diet, lifestyle instructions according guidelines.

INTERVENTIONS:
Behavioral: therapeutic monitoring — According to the glucose lever recorded by FreeStyle Libre H (Flash Continuous Glucose Monitoring System) ,the investigators give the intervention group instructions to adjust their diet and lifestyle to abtain a good glucose control.
  Arms: therapeutic monitoring

SUMMARY:
The purpose of this study is to conduct a multicenter prospective randomized controlled clinical trial, evaluating the effects of "therapeutic monitoring" on blood glucose control in type 2 diabetes.

DETAILED DESCRIPTION:
In our study, about 480 type 2 diabetes patients will be enrolled from multiple centers in China. All participants will be randomly assigned into either the intervention group or the control group. All patients will be given basic diet, lifestyle instruction according to guidelines from home and abroad. The intervention group will be instructed to adjust the diet according to the ambulatory glucose profile (AGP) and the recorde log monitored by the continuous glucose monitoring system, thereby implementing "therapeutic monitoring". All patients will maintain the drug treatment unchanged and make the glucose level as far as possible within the target range (>3.9 and ≤10mmol/L), and record the amount of various food, then maintain the dietary pattern and the amount unchanged until the end of the study.

The primary objective is to evaluate the effects of "therapeutic monitoring" on blood glucose control in type 2 diabetes, as measured by change in HbA1c level from baseline to 12-week follow-up in both intervention group and control group.

THe secondary endpoint are 1) 1)Difference in TIR (time in range, time in target glucose range, 3.9-10.0mmol/L) at 12 weeks in both groups. 2)Fasting plasma glucose (FPG), lipids and other metabolic related components and parameters such as BMI will be measured. 3)Using questionnaires to evaluate the patients' satisfaction with Flash Glucose Monitoring System.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes defined as WHO(1999) diagnostic criteria;
* HbA1c ≥ 7% and ≤ 9% at screening; and fasting plasma glucose ≥ 7.0mmol/L, and <13.3mmol/L;
* Duration: 3 months~15 years;
* BMI: 24~ 28 kg/m2;
* Using 1-3 oral medications when enrolled, and the treatment pattern was stable for at least 3 months and can maintain during this study period;
* Sign the informed consent. Details please see the study protocol.

Exclusion Criteria:

* There are serious diabetic complications, heart, brain, liver and kidney diseases, allergic diseases and organic diseases;
* The subject is currently pregnant, intends to become pregnant or is unwilling or unable to contraception during the study (female only);
* The subject has symptoms or signs of skin lesions, scab, redness, infection or edema at the sensor application site that may affect the accuracy of sensor application or interstitial glucose measurements;
* The subject has a concomitant disease and the investigator believes it will affect the study or pose a risk to the safety or benefit of the subject or research worker.
* An X-ray, MRI, or CT examination is scheduled during the study period, and the appointment could not be changed to before the study started or after the study ended;
* Take aspirin > 200 mg / day, and the drug may be added during the entire study period; Details please see the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2019-12-10 (Estimated); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-11-15 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 12 weeks
  Analysis the difference in HbA1c between intervention and control groups at 12 weeks

SECONDARY OUTCOMES:
TIR | 12 weeks
  time in range, time in target glucose range, 3.9-10.0mmol/L
Fasting glucose levels | 12 weeks
  Analysis the difference in Fasting glucose levels between intervention and control groups at 12 weeks
Fasting c-peptide levels | 12 weeks
  Analysis the difference in Fasting c-peptide levels between intervention and control groups at 12 weeks
Serum Triglycerides | 12 weeks
  Analysis the difference in Serum Triglycerides levels between intervention and control groups at 12 weeks
Serum total Cholesterol | 12 weeks
  Analysis the difference in Serum total Cholesterol levels between intervention and control groups at 12 weeks
Serum HDL-c | 12 weeks
  Analysis the difference in Serum HDL-c levels between intervention and control groups at 12 weeks
Serum LDL-c | 12 weeks
  Analysis the difference in Serum LDL-c levels between intervention and control groups at 12 weeks
Body weight | 12 weeks
  weight in kilograms
Height | 12 weeks
  height in meters
Blood pressure | 12 weeks
  analyses the difference of blood pressure in both groups
Creatinine | 12 weeks
  analyses the difference of Creatinine in both groups
Uric acid | 12 weeks
  analyses the difference of Uric acid in both groups
UCAR | 12 weeks
  Analysis the difference in Urinary albumin creatinine ratio（UCAR） between intervention and control groups at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Weiqing Wang, MD,PHD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China